CLINICAL TRIAL: NCT06070090
Title: Tapping in Together: A Pilot Study on Group Acupuncture for Ketamine Experience Integration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Oriental Medicine Austin (Other)
Responsible Party: Principal Investigator, Marjorie Navarro, Licensed Acupuncturist, Academy of Oriental Medicine Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23C.MN
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acupuncture
Keywords: Ketamine
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: An intention-to-treat approach will be used to approximate real-world conditions wherein results will be included even if a participant decides not to participate in the group acupuncture session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This is the group of participants who will receive group acupuncture after a ketamine experience.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — The traditional East Asian methods of treating disease by inserting needles along specific pathways or meridians.
  Other Names: Acupuncture Therapy

SUMMARY:
The goal of this pilot trial is to learn about using acupuncture for ketamine experience integration in adults aged 21-65 who are medically cleared for a ketamine prescription. The aim is to inform future controlled trials investigating efficacy by evaluating the success of:

* recruitment
* retention
* assessment procedures
* implementation of group acupuncture interventions performed just after a ketamine experience

Participants will be given acupuncture in a group setting after a small-group ketamine experience. The following day, participants will be asked to complete a few brief surveys about their experience.

DETAILED DESCRIPTION:
The study will solicit participants to enroll in a physician-supervised ketamine experience directly followed by group acupuncture administered in New York City, between October 1, 2023 and February 28, 2024. A group of 12-28 participants will be enrolled in the study and assigned a participant ID once screened by the researcher and medically approved by the prescribing physician.

Group acupuncture treatments will be conducted one hour after a group ketamine experience commences. The group acupuncture sessions will start with the researcher approaching each participant individually and asking to examine their pulse and tongue. The participants will be given an opportunity to share any information they would like to about specific issues they would like to address with acupuncture. If nothing is shared, the researcher will select treatment points based on their pulse, tongue, body palpation, and intake data. The general location of the points selected will be shared with the participant to gain their consent for treating those areas prior to needle insertion. While the acupuncture needles are retained, participants will rest with music playing. The needles will then be removed, one at a time, from each patient in order of treatment (unless a participant requests needle removal before then). After needle removal, the participants will be asked to sit up for a few minutes before exiting the treatment room. Both the licensed acupuncturist researcher and a psychotherapist will be in the treatment room throughout the 1-hour group acupuncture session.

Participants will be emailed a validated survey via a REDCap secure link before the group acupuncture session (if they had a previous ketamine experience), after their group acupuncture session as well as 3 months from the date of their group acupuncture session. Participants will also be sent optional feedback forms through REDCap after each acupuncture session.

ELIGIBILITY:
Inclusion Criteria:

* between ages 21-65
* participant in a group ketamine experience between October 1, 2023 and February 28, 2024

Exclusion Criteria:

* currently pregnant or breastfeeding
* has a terminal illness
* does not pass medical clearance for ketamine prescription

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Experienced Integration Scale (EIS) | One day after experience
  The scale is intended to gain a sense of the status of a participant's integration process after a psychedelic experience. Participants are asked to rate their agreement to 12 statements using a five-point Likert scale with the anchors "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree." The items are worded in a positive direction, so that higher scores indicating greater integration.
Experienced Integration Scale (EIS) | Three months after experience
  The scale is intended to gain a sense of the status of a participant's integration process after a psychedelic experience. Participants are asked to rate their agreement to 12 statements using a five-point Likert scale with the anchors "strongly disagree," "disagree," "neither agree nor disagree," "agree," and "strongly agree." The items are worded in a positive direction, so that higher scores indicating greater integration.

CONTACTS AND LOCATIONS:
Overall Officials: William Morris, PhD, DAOM, Study Chair — Academy of Oriental Medicine Austin
Locations (1):
- Cardea Ketamine Space, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No